CLINICAL TRIAL: NCT02660489
Title: Effect of the CRTH2 Antagonist OC459 on the Response to Rhinovirus Challenge in Asthma
Brief Title: Effect of OC459 on the Response to Rhinovirus Challenge in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Atopix Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORCA2015
Record Dates: First submitted 2016-01-12; First posted 2016-01-21 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Asthma; Rhinovirus; Picornaviridae Infections; Common Cold
Keywords: CRTH2 antagonist; Prostaglandin D2 receptor; Anti-Asthmatic Agents; OC459; Allergic asthma; Eosinophilia
MeSH Terms: conditions — Asthma; Picornaviridae Infections; Common Cold; Eosinophilia | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OC459 (CRTH2 antagonist) (Experimental): OC459 50mg once daily for 5 weeks
  Interventions: Drug: OC459; Other: Rhinovirus
- Placebo (Placebo Comparator): Placebo tablet once daily for 5 weeks
  Interventions: Drug: Placebo; Other: Rhinovirus

INTERVENTIONS:
Drug: OC459
  Other Names: OC000459
  Arms: OC459 (CRTH2 antagonist)
Drug: Placebo
  Arms: Placebo
Other: Rhinovirus — Inoculation with rhinovirus serotype 16

SUMMARY:
The aim of this study is to assess the effectiveness of a CRTH2 receptor antagonist, OC459, in preventing or attenuating the worsening of asthma symptoms during rhinovirus infection. The study is a double blind, randomised trial in which half the subjects will receive OC459 and the other half placebo, before being inoculated with rhinovirus, that would normally induce a worsening of asthma symptoms i.e. an exacerbation.

DETAILED DESCRIPTION:
Asthma is the most common chronic respiratory disease, and in many countries prevalence is rising. The major morbidity, mortality and health care costs related to asthma are a result of periods of acutely increased symptomatology called 'exacerbations'. Most exacerbations are caused by rhinovirus, the virus associated with the common cold. There are few treatments to prevent and treat exacerbations, and despite these >50% of adult asthmatics reported having an exacerbation in the last year. There is therefore a major unmet need.

Experimentally inoculating patients with asthma with rhinovirus, a methodology that has been safely used for >15 years, induces an infection and worsening symptoms in ~85%. This model offers the possibility to investigate treatment effects on asthma exacerbations with a small number of subjects, minimising the numbers exposed to a novel drug with limited safety data. In contrast, trials of therapies powered to evaluate an effect on naturally occurring exacerbations require several hundred subjects, a long study period to capture enough events, and are significantly more expensive to carry out.

Using this model the investigators have shown that several inflammatory molecules, including prostaglandin D2 (PGD2), are significantly increased during rhinovirus-induced asthma exacerbations, with the levels of PGD2 strongly correlating with the severity of the symptoms. Moreover other studies have shown that when PGD2 binds the CRTH2 receptor, it stimulates the release of a number of inflammatory molecules also associated with asthma exacerbations. Blocking the CRTH2 receptor therefore appears an extremely promising target with potential to limit the virus-induced inflammation underpinning many asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18--55 years
* Male or female
* Clinical diagnosis of asthma for at least 6 months prior to screening
* An Asthma Control Questionnaire (ACQ) Score >0.75
* Positive histamine challenge test (PC20 <8 µg/ml, or <12 µg/ml and bronchodilator response ≥ 12%)
* Worsening asthma symptoms with infection since last change in asthma therapy
* Positive skin prick test to common aeroallergens (e.g. animal epithelia, dust mite)
* Treatment comprising inhaled corticosteroids (ICS) or combination inhaler (Long -Acting Beta Agonist with ICS), with a daily ICS dose of at least 100mcg fluticasone or equivalent.
* Participant is willing for their GP to be informed of their participation.
* English speaker

Exclusion Criteria:

* Presence of clinically significant diseases other than asthma, which, in the opinion of the investigator, may either put the patient at risk because of participation in the trial, or diseases which may influence the results of the study or the patient's ability to take part in it
* Smoking history over past 12 months
* Seasonal allergic rhinitis symptoms at screening
* Asthma exacerbation or viral illness within the previous 6 weeks
* Current or concomitant use of oral steroids, anti--leukotrienes or monoclonal antibodies
* Pregnant or breast-feeding women (patients should not be enrolled if they plan to become pregnant during the time of study participation)
* Contact with infants <6 months or immunocompromised persons, elderly and infirm at home or at work
* Subjects who have known evidence of lack of adherence to medications and/or ability to follow physician's recommendations

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian L Johnston, MBBS PhD, Principal Investigator — National Heart & Lung Institute, Imperial College London
Locations (1):
- St Mary's Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Started | 22 | 22
Completed | 16 (Completed with confirmed rhinovirus infection) | 14 (Completed with confirmed rhinovirus infection)
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 3
Not completed — no rhinovirus infection | 4 | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed the study and had confirmed rhinovirus infection
Groups:
- Total: Total of all reporting groups
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (8.9) | 25.4 (3.8) | 25.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Lower Respiratory Symptom Score
Description: Sum of daily scores for 14 days. Seven symptoms (cough on waking, wheeze on waking, daytime cough, daytime wheeze, daytime chest tightness, daytime breathlessness, nocturnal cough/wheeze/breathlessness) ranked from 0 (none) to 3 (severe). Range 0 to 294; higher is more symptomatic.
Time Frame: During 14 days following rhinovirus inoculation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
score on a scale | 21 [13.3 to 46.5] | 18 [9.8 to 51.5]
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Asthma Control Questionnaire (ACQ)-6 Score
Description: Change from baseline (rhinovirus inoculation, day 0) to day 10. The ACQ was developed to measure the adequacy of asthma control in clinical research and in clinical practice. The ACQ-6 asks subjects to grade their asthma control, assessed through six questions, over the previous seven days. Each question is rated on a seven-point scale ranging from 0 (well controlled) to six (extremely poorly controlled). The ACQ-6 score is the mean of the scores on the 6 items. Mean scores of =<0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma.
Time Frame: Baseline, 10 days post rhinovirus inoculation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
score on a scale | -0.01 (0.68) | 0.17 (0.71)
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.49, t-test, 2 sided

3. Secondary Outcome: Percentage Change in Peak Expiratory Flow Rate
Description: Percentage change from baseline (rhinovirus inoculation, day 0) to trough during infection (up to day 14)
Time Frame: Baseline and up to 14 days post rhinovirus inoculation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
percentage change | -16.9 (10.2) | -13.1 (12.8)
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.50, t-test, 2 sided

4. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Percentage change from baseline (rhinovirus inoculation, day 0) to trough during infection (up to day 14)
Time Frame: Baseline and up to 14 days post rhinovirus inoculation
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
percentage change | -18.5 (11.3) | -12.7 (14.0)
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.36, t-test, 2 sided

5. Secondary Outcome: Change in Exhaled Nitric Oxide (FeNO)
Description: Percentage change from baseline (rhinovirus inoculation, day 0) to peak during infection (highest of measurements on days 3, 5, 7, 10 post inoculation)
Time Frame: Baseline and up to 10 days post rhinovirus inoculation
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
percentage change | 58 [27 to 101] | 23 [0 to 77]
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Changes in Airway Hyper Responsiveness (Histamine)
Description: Assessed as the provocation concentration of histamine producing a 20% fall in FEV1, or PC20 Change from baseline (rhinovirus inoculation, day 0) to day 7
Time Frame: Baseline and 7 days post rhinovirus inoculation
Population: Two subjects (one from each group) were unable to complete PC20 at one of the time points for logistical reasons
Measure: Median (Inter-Quartile Range); unit: mg/mL
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 15 | 13
mg/mL | -0.1 [-0.77 to 0.21] | -0.64 [-2.19 to -0.31]
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Viral Load (in Nasal Lavage Samples)
Description: Peak during infection (up to day 14)
Time Frame: Up to 14 days post rhinovirus inoculation
Measure: Median (Full Range); unit: viral copies / mL
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
viral copies / mL | 445861 [0 to 9025667] | 215782 [0 to 25240371]
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.75, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Total Upper Respiratory Symptom Score
Description: Sum of daily scores for 14 days. Eight upper respiratory symptoms (sneezing; runny nose; blocked or stuffy nose; sore throat or hoarse voice; headache or face pain; generally unwell; chill, fever or shivery; cough) ranked from 0 (none) to 3 (severe). Range 0 to 336; higher is more symptomatic.
Time Frame: During 14 days following rhinovirus inoculation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
Number analyzed (Participants) | 16 | 14
score on a scale | 33 [20.5 to 63.3] | 41 [18.5 to 63.8]
Statistical Analysis 1: Comparison: OC459 (CRTH2 Antagonist) vs Placebo; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 9 weeks
Description: Participants were asked to record adverse events in a study diary that was completed daily.
  Participants were also asked about adverse events at study visits.
Arm/Group | OC459 (CRTH2 Antagonist) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OC459 (CRTH2 Antagonist) (N=22) | Placebo (N=22)
Headache (Nervous system disorders) | 4 (17) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT02660489/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT02660489/SAP_001.pdf